CLINICAL TRIAL: NCT04176068
Title: Combined Focused Ultrasound and Calcium Hydroxylapatitie Filler for Skin Laxity
Brief Title: Combined Focused Ultrasound and Calcium Hydroxylapatitie Filler for Skin Laxity and Volume Restoration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Vice Chair of Clinical Research, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20184856
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Combined microfocused ultrasound and calcium hydroxylapatite (Experimental): One-time intense microfocused ultrasound with calcium hydroxylapatite injection to one anterior lower thigh with option for additional filler injection at 6 weeks, 12 weeks, and 24 weeks. Optional combined treatment of the opposite lower anterior thigh at week 24 with no further follow up.
  Interventions: Combination Product: calcium hydroxylapatite (Radiesse) and IFUS (Ulthera)

INTERVENTIONS:
Combination Product: calcium hydroxylapatite (Radiesse) and IFUS (Ulthera) — Patients will receive IFUS to a randomly chosen side. Immediately after IFUS treatment, patients will receive the first CaHA injection. Injections will be given in the lower, anterior third of the thigh, above the knee. Only dermatology faculty will perform the filler injections. The patients will be instructed to return to the office in 6 weeks, 12 weeks, and 24 weeks (+/- 5 business days) for their next appointment for follow-up and injection of CaHA if deemed necessary by the investigator. At all visits (Visits 1-4) patients will have photographs and unblinded physician/patient questionnaires will be completed. At Visit 4 (24 weeks +/- 5 business days), patients will be given the option to receive treatment for skin laxity to the previously untreated side. If the patient chooses to receive treatment, patients will receive their second IFUS and CaHA combination treatment at this time. They will not receive further treatment after this visit.
  Other Names: intense microfocused ultrasound

SUMMARY:
Non-invasive treatment options such as focused ultrasound has been used with success for the treatment of skin laxity in various parts of the body including the face, neck, décolletage, arms, buttocks, thighs, and legs. With the increasing demand for greater results, researchers have started combining modalities together such as focused ultrasound and intradermal filler, with promising effects for skin laxity and volume restoration. This study aims to elucidate the efficacy and added benefits of a combination therapy using focused ultrasound (Ulthera) and calcium hydroxylapatite (Radiesse) for the treatment of skin laxity and volume restoration of the lower thighs, specifically the lower anterior third of the thigh.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibit skin aging and laxity that will benefit from treatment as determined by the investigator/physician.
2. Subjects between the ages of 18-85 years old, at the time of consent.
3. Subjects may be male or female.
4. Subjects can be of any Fitzpatrick Skin type (I-VI).
5. Subjects must be able and willing to give written informed consent and to comply with the requirements of this protocol. The consent form has been standardized in English. For those patients who do not read and understand English, a consent form will be standardized and provided in a language that they read and understand.

Exclusion Criteria:

1. Children and adolescents (less than 18 years old).
2. Subjects who are not willing or able to provide written consent.
3. Individuals with any significant medical history including skin disorders and eating disorders as determined by the investigator/physician.
4. Subjects on any substances affecting blood coagulation (including but not limited to aspirin and other non-steroid anti-inflammatory drugs, warfarin, vitamin E, fish oil, heparin, low-molecular weight heparin, novel anti-coagulants).
5. Subjects with known blood coagulopathies.
6. Subjects with a compromise of local blood supply (including but not limited to recent surgery, severe scarring, autoimmune diseases involving the lower thigh such as lupus, morphea, sarcoid or mixed connective tissue disease).
7. Subjects who have received any treatment for skin laxity or liposuction in the last 12 weeks.
8. Subjects who have experienced an increase or decrease in body weight of more than 10% in the past 24 weeks.
9. Subjects who have a known hypersensitivity reaction to calcium hydroxylapatite or the components of the filler product.
10. Subjects with open wounds in the area of ultrasound treatment.
11. Subjects with pacemakers and/or electronic device implants in the area of ultrasound treatment.
12. Female patients who are planning a pregnancy, currently pregnant or nursing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of combined therapy at 12 weeks | 12 weeks
  To determine the efficacy of intense focused ultrasound (IFUS) + calcium hydroxylapatite (CaHA) filler for the correction of skin laxity of the lower thigh as assessed by a blinded and an unblinded physician Global Aesthetic Improvement Scale (scale 1-7 with 1 being much improved and 7 being much worse) at 12 weeks.

SECONDARY OUTCOMES:
Efficacy of combined therapy at 24 weeks | 24 weeks
  To determine the efficacy of IFUS and CaHA filler for the correction of skin laxity of the lower thigh as assessed by a blinded and an unblinded physician Global Aesthetic Improvement Scale (scale 1-7 with 1 being much improved and 7 being much worse) at 24 weeks.
Efficacy with Merz Aesthetic scale at 12 and 24 weeks | 24 weeks
  To determine the efficacy of IFUS and CaHA filler for the correction of skin laxity of the lower thigh as assessed by a blinded and an unblinded physician Merz Aesthetic Scale (Grade 0-4 with 0 being no skin laxity and 4 being very severe skin laxity) at 12 and 24 weeks.
Patient satisfaction at 24 weeks | 24 weeks
  To determine patient satisfaction 24 weeks post-treatment of IFUS + CaHA for the treatment of skin laxity of the lower thigh as assessed on a scale of 0-10 (with 0 being not satisfied and 10 being very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Mesinkovska, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Dermatology Clinical Research Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No